CLINICAL TRIAL: NCT05041712
Title: Biomarkers of Brain Injury in Critically-Ill Children on Extracorporeal Membrane Oxygenation
Acronym: BEAM
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00215794; 1R01NS106292 (NIH)
Record Dates: First submitted 2021-08-10; First posted 2021-09-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Extracorporeal Membrane Oxygenation; Children; Neurologic Injury
Keywords: Brain Injury Biomarkers; Neurodevelopmental Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and ultrafiltrate fluid (if the participant is on renal replacement therapy or ultrafiltration) will be collected daily on ECMO days #1-5, then every 3 days thereafter while on ECMO.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case cohort: Observational study of children between the ages of 2 days to < 18 years who are cannulated onto ECMO at participating sites
- Control cohort: Observational study of children between the ages of 2 days to < 18 years admitted to the Johns Hopkins Pediatric Intensive Care Unit (PICU) or Pediatric Cardiac Intensive Care Unit (PCICU) for any reason.

SUMMARY:
The BEAM study is a multicenter, prospective, observational study in children supported on extracorporeal membrane oxygenation (ECMO). The primary goals of this study are to develop and refine a brain injury multimarker panel for accurate neurologic monitoring at the bedside and early classification of mortality and disability outcomes of critically ill children supported on ECMO.

DETAILED DESCRIPTION:
The specific aims are to:

1. Determine if circulating levels of brain injury markers during ECMO and brain MRI abnormalities within 6 weeks after ECMO are associated with survival at 18 months after ECMO with a score ≥85 on the Vineland Adaptive Behavior Scales, third edition (VABS-III).
2. Determine whether the presence and degree of inflammation during ECMO and markers of neuroinflammation on brain magnetic resonance spectroscopy (MRS) within 6 weeks after ECMO are associated with survival at 18 months after ECMO with a score ≥85 on VABS-III.
3. Determine whether metabolic and lipid neuroinflammatory pathways will distinguish between at-risk for, acute, and recovery phases of neurologic injury (NI) during ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Children (2 days to <18 years) cannulated onto ECMO and admitted to a pediatric or cardiac Intensive Care Unit at participating institutions.

Exclusion Criteria:

* ECMO cannulation at an outside institution with transport to a study site >24 hours after ECMO initiation
* Limitation of care (e.g., family planning to withdraw support)
* Brain death evaluation within 24 hours of ECMO cannulation
* Inability to speak or understand English or Spanish
* Pregnancy.

Ages: 2 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 225 children who are cannulated onto ECMO and admitted to a pediatric or cardiac Intensive Care Unit at participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Change in Vineland Adaptive Behavior Scales-Third Edition (VABS-3) | Baseline and 18 months post-ECMO
  VABS-3 is a 381-item caregiver report measure that was developed to assess adaptive behavior. The questionnaire is divided into 4 domains of adaptive behavior: 1) communication, 2) daily living, 3) social skills and relationships, and 4) physical activity. Each item is rated 0 (never), 1 (sometimes), or 2 (usually or often) as how often the child does the behavior independently without help or reminders. The overall adaptive composite score has a mean of 100 and standard deviation of 15 with lower scores indicating worse intellectual disability.

SECONDARY OUTCOMES:
Change in Functional Status Scale (FSS) | Baseline and at hospital discharge, up to 18 months post-ECMO
  The FSS examines 6 domains of functioning: 1) mental status; 2) sensory; 3) communication; 4) motor function; 5) feeding; and 6) respiratory and each domain receives a score of 1 (normal), 2 (mild dysfunction), 3 (moderate dysfunction), 4 (severe dysfunction), or 5 (very severe dysfunction). Final scores range from 6 to 30 with higher scores indicating greater dysfunction.
Change in Pediatric Cerebral Performance Category (PCPC) | Baseline and at hospital discharge, up to 18 months post-ECMO
  PCPC consists of a 6-point scale: 1) normal; 2) mild disability; 3) moderate disability; 4) severe disability; 5) coma/vegetative state; 6) brain death. Higher scores indicating worse performance or functional morbidity
Change in Pediatric Overall Performance Category (POPC) | Baseline and at hospital discharge, up to 18 months post-ECMO
  POPC consists of a 6-point scale: 1) good overall performance; 2) mild overall disability; 3) moderate overall disability; 4) severe overall disability; 5) coma/vegetative state; 6) brain death. Higher scores indicating worse performance or functional morbidity
Change in Pediatric Quality of Life (PedsQL) Inventory | Baseline and 18 months post-ECMO
  The PedsQL Inventory is a 36-item (for infants 1-12 months), 45 item (for infants 13-24 months) or 23-item (children 2-18) questionnaire with established validity and reliability for health outcomes measurements in pediatric populations, including former PICU patients. The PedsQL is used as a parent proxy report for all ages, as well as self-report in children between 5 and 18 years. The scales are divided into 4 domains of functioning: 1) physical functioning, 2) emotional functioning, 3) social functioning and either 4) cognitive functioning (on the infant scales) or school functioning (on the child scales). Each item on the parent proxy report receives a score of 0 (never), 1 (almost never), 2 (sometimes), 3 (often), or 4 (almost always). Each score on the child report receives a score of 0 (not at all), 2 (sometimes), or 4 (a lot). Final transformed scores range from 0-100 with higher scores indicating better health-related quality of life.
Consumer Assessment of Healthcare Providers and Systems (CAHPS) Child Survey 5.0H with the Children with Chronic Conditions (CCC) Item Set | 18 months post-ECMO
  The CAHPS CCC is an 81-item questionnaire that provides information on parents' experiences with their child's health care and gives a general indication of how well the health care meets their expectations. Five CCC-specific results are calculated for each population: 1) access to specialized services, 2) family-centered care: personal doctor who knows the child, 3) coordination of care for children with chronic conditions, 4) access to prescription medication, and 5) family-centered care: getting needed information.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Bembea, MD, MPH, PhD, Principal Investigator — Johns Hopkins University
Locations (11):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided